CLINICAL TRIAL: NCT03714178
Title: PEFCAT: A Safety and Feasibility Study of the FARAPULSE Endocardial Ablation System to Treat Paroxysmal Atrial Fibrillation
Brief Title: A Safety and Feasibility Study of the FARAPULSE Endocardial Ablation System to Treat Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0267
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients undergoing catheter ablation of paroxysmal atrial fibrillation and meeting all protocol inclusion/exclusion criteria will be treated with the FARAPULSE Endocardial Ablation System.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- FARAPULSE Endocardial Ablation (Experimental): Subjects who are treated with the FARAPULSE Endocardial Ablation System for paroxysmal atrial fibrillation.
  Interventions: Device: FARAPULSE Endocardial Ablation System

INTERVENTIONS:
Device: FARAPULSE Endocardial Ablation System — Endocardial ablation using the FARAPULSE Endocardial Ablation System.

SUMMARY:
PEFCAT is a prospective, single-arm, multi-center, safety and feasibility study evaluating the FARAPULSE Endocardial Ablation System for the treatment of paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
Patients undergoing catheter ablation for paroxysmal atrial fibrillation will be screened for enrollment per protocol inclusion and exclusion criteria. Enrolled patients will then undergo ablation using the FARAPULSE Endocardial Ablation System. Subjects will be followed at 7 days, 30 days, 75 days, 6 months, and 12 months with a blanking period for recurrent atrial fibrillation or atrial tachycardia of 3 months following the PEF (pulsed electric field) catheter ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented drug resistant symptomatic PAF who have:

   1. Confirmed AF: Documentation may include ECG, transtelephonic monitor (TTM), Holter monitor, implanted devices, telemetry strip or similar, recorded within one year prior to enrollment and showing at least 30 seconds of AF.
   2. Frequent AF, defined as ≥ 2 episodes within 6 months of enrollment.
   3. Failed AFD, meaning therapeutic failure of at least one antiarrhythmic drug (AFD; class I - IV) for efficacy and / or intolerance
2. Patients who are ≥ 18 and ≤ 75 years of age on the day of enrollment.
3. Patient participation requirements:

   1. Lives locally
   2. Is willing and capable of providing Informed Consent to undergo study procedures
   3. Is willing to participate in all examinations and follow-up visits and tests associated with this clinical study.

Exclusion Criteria:

1. Use of amiodarone within 3 months prior to enrollment
2. Atrial fibrillation that is any of the following

   1. Persistent (by diagnosis or duration > 7 days)
   2. Secondary to electrolyte imbalance, thyroid disease, alcohol abuse or other reversible / non-cardiac causes
   3. Requires ≥ 3 cardioversions in the preceding 12 months
3. Cardiac anatomical exclusions by imaging within 3 months prior to enrollment:

   1. Left atrial anteroposterior diameter ≥ 5.0 cm as documented by transthoracic echocardiography (TTE) or computed tomography (CT)
   2. Left ventricular ejection fraction ≤ 40% as documented by TTE
4. Any of the following cardiac procedures, implants or conditions:

   1. Clinically significant arrhythmias other than AF
   2. Hemodynamically significant valvular disease
   3. Prosthetic heart valve
   4. NYHA Class III or IV CHF
   5. Previous endocardial or epicardial ablation or surgery for AF
   6. Atrial or ventricular septal defect closure
   7. Atrial myxoma
   8. Left atrial appendage device or occlusion
   9. Pacemaker, ICD or CRT
   10. Significant or symptomatic hypotension
   11. Bradycardia or chronotropic incompetence
   12. History of pericarditis
   13. History of rheumatic fever
5. Any of the following within 3 months of enrollment:

   1. Myocardial infarction
   2. Unstable angina
   3. Percutaneous coronary intervention
   4. Heart surgery including coronary artery bypass grafting
   5. Heart failure hospitalization
   6. Stroke or TIA
   7. Clinically significant bleeding
   8. Pericarditis or pericardial effusion
   9. Left atrial thrombus
6. History of blood clotting or bleeding abnormalities.
7. Contraindication to, or unwillingness to use, systemic anticoagulation
8. Contraindications to CT or MRI
9. Sensitivity to contrast media not controlled by premedication
10. Women of childbearing potential who are pregnant, lactating or not using birth control
11. Serious or untreated medical conditions that would prevent participation in the study, interfere with assessment or therapy, or confound data or its interpretation, including but not limited to

    1. Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
    2. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or significant dyspnea
    3. Chronic renal insufficiency of < 60 mL/min/1.73 m2, any history of renal dialysis, or history of renal transplant
    4. Active malignancy or history of treated cancer within 24 months of enrollment
    5. Clinically significant gastrointestinal problems involving the esophagus, stomach and/or untreated acid reflux
    6. Clinically significant infection
    7. Predicted life expectancy less than one year
12. Clinically significant psychological condition that in the investigator's opinion would prohibit the subject's ability to meet the protocol requirements
13. Current or anticipated enrollment in any other clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, PhD, Principal Investigator — Nemocnice Na Homolce
Locations (2):
- Nemocnice Na Homolce, Prague, Czechia
- CHU Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reddy VY, Neuzil P, Koruth JS, Petru J, Funosako M, Cochet H, Sediva L, Chovanec M, Dukkipati SR, Jais P. Pulsed Field Ablation for Pulmonary Vein Isolation in Atrial Fibrillation. J Am Coll Cardiol. 2019 Jul 23;74(3):315-326. doi: 10.1016/j.jacc.2019.04.021. Epub 2019 May 11. PMID 31085321

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FARAPULSE Endocardial Ablation
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FARAPULSE Endocardial Ablation
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Czechia | 50
  France | 21
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.3 (4.4)
Left atrial diameter [Mean (Standard Deviation); unit: cm] | 4.1 (0.5)
Atrial Fibrillation history (number of months) [Mean (Standard Deviation); unit: months] | 16.61 (23.94)
LVEF % [Mean (Standard Deviation); unit: percentage of left ventricular ejection] | 62.1 (6.3)
CHA2DS2VASC [Mean (Standard Deviation); unit: units on a scale] — Tool used to predict the risk of ischemic stroke in patients with AF, which can help guide the decision to treat those patients with anticoagulants. Calculated by adding the number of risk factors.CHF,hypertension,age≥75diabetesstroke/TIA/TE, vascular disease, age 65-74 years & sex. Each risk factor adds a point to the risk score, except for Age ≥ 75 years & Stroke/TIA/TE, which both add 2 pointsscore of 0 represents a patient having no additional risk factors. The ESC guidelines considers a score of 1 to be moderate risk and a score ≥ 2 to be high risk. Range: 0 (lower risk) - 9 (higher risk)
  units on a scale | 1.8 (1.6)
Patient that failed any AntiArrhythmic Drugs [Count of Participants; unit: Participants] | 69
Smoking [Count of Participants; unit: Participants] | 38
Dyslipidemia [Count of Participants; unit: Participants] | 24
COPD [Count of Participants; unit: Participants] | 1
PPM/ICD [Count of Participants; unit: Participants] | 0
Unstable angina [Count of Participants; unit: Participants] | 0
NYHA Heart Failure Class I [Count of Participants; unit: Participants] — I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants | 18
NYHA Heart Failure Class II [Count of Participants; unit: Participants] — I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants | 3
NYHA Heart Failure Class III [Count of Participants; unit: Participants] — I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants | 0
NYHA Heart Failure Class IV [Count of Participants; unit: Participants] — I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants | 0
Any History of Structural heart disease [Count of Participants; unit: Participants] | 3
Cerebrovascular disease [Count of Participants; unit: Participants] | 6
Cardiac Surgery [Count of Participants; unit: Participants] | 2
Diabetes [Count of Participants; unit: Participants] | 7
Hypertension [Count of Participants; unit: Participants] | 42
Hyperthyroidism [Count of Participants; unit: Participants] | 3
Hypothyroidism [Count of Participants; unit: Participants] | 9
Myocardial infarction [Count of Participants; unit: Participants] | 3
Peripheral vascular disease [Count of Participants; unit: Participants] | 3
Pulmonary hypertension [Count of Participants; unit: Participants] | 0
Renal dysfunction/failure [Count of Participants; unit: Participants] | 1
Sleep apnea [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint for This Study is the Composite Safety Endpoint (CSE) Defined as the Proportion of Patients With Early-onset and Late-onset Serious Adverse Events (SAEs) Which Are Device- or Procedure-related.
Description: Early onset (within 30 days of any endocardial ablation for atrial fibrillation). Occurrence of any one of the below events will qualify a subject as a safety failure.
  * Death
  * Myocardial infarction (MI)
  * Persistent diaphragmatic paralysis
  * Stroke or transient ischemic attack (TIA)
  * Peripheral or organ thromboembolism
  * Pericarditis
  * Cardiac tamponade / perforation
  * Vascular access complications
  * Hospitalization (initial or prolonged)*
  * Heart block
    * Late onset (any time during follow-up)
  * Pulmonary vein (PV) stenosis (> 70% diameter reduction from baseline)
  * Atrio-esophageal fistula * Excludes hospitalization (initial & prolonged) solely due to arrhythmia (AF/Atrial Flutter/Atrial Tachycardia) recurrence or due to non-urgent cardioversion (pharmacological or electrical).
Time Frame: 30 days~12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE Endocardial Ablation
Number analyzed (Participants) | 71
Participants | 2

2. Secondary Outcome: Feasibility: Pulmonary Vein Isolation
Description: The proportion of subjects that achieve Acute Procedural Success (APS) defined as the percutaneous endocardial creation of a complete, electrically isolating set of lesions around the ostia of the pulmonary veins (PVI) using the FARAPULSE Endocardial Ablation System during the first procedure, as clinically assessed by entrance and/or exit block performed ≥ 20 minutes after the last PVI lesion is made.
Time Frame: 1 Day (Acute)
Measure: Number; unit: Proportion of participants
Arm/Group | FARAPULSE Endocardial Ablation
Number analyzed (Participants) | 71
Proportion of participants | 1.0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | FARAPULSE Endocardial Ablation
All-Cause Mortality (participants affected / at risk) | 0/71
Serious Adverse Events (participants affected / at risk) | 11/71
Other Adverse Events (participants affected / at risk) | 17/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Endocardial Ablation (N=71)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Air Embolism (Vascular disorders) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 2 (2)
Inguinal Hernia (Gastrointestinal disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardioversion (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Endocardial Ablation (N=71)
Chronic Gastritis (Gastrointestinal disorders) | 9
Oedema peripheral (General disorders) | 4 (71)
Palpitations (Cardiac disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT03714178/Prot_SAP_000.pdf